CLINICAL TRIAL: NCT03258450
Title: The Feasibility and Acceptability of a Psychosocial Intervention for Advanced Colorectal Cancer Patients
Brief Title: Effectiveness of a Psychosocial Intervention for Colorectal Cancer
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Principal Investigator, Irene Teo, Clinical Psychologist , Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSRNIG
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psycho-behavioural intervention arm (PBI) (Experimental): Participants will receive 4 sessions(PBI) that lasts approximately 60 mins.
  Interventions: Behavioral: Psycho-behavioural intervention arm (PBI)
- Waitlist Control Arm (WLC) (No Intervention): The WLC group receives standard usual care before being offered the same PBI protocol and assessment thereafter.

INTERVENTIONS:
Behavioral: Psycho-behavioural intervention arm (PBI) — The first session introduces the rationale of the intervention and is designed to encourage participants to recognize the autonomous role they can play in their health and well-being. Patients will be trained on breathing as a relaxation technique. The second session focuses on building behavioural skills to manage common symptoms for colorectal cancer patients. The third session focuses on cognitive strategies to address worries and existential distress. The last session focuses on maximizing social support and applying skills learned so far in dealing with loved ones. Participants will be provided an MP3 player that contains the relaxation exercise recording and a folder with summaries of the session content.
  Arms: Psycho-behavioural intervention arm (PBI)

SUMMARY:
Studies have reported about one-third to half of advanced cancer patients experience psychological distress yet the mental healthcare needs of these patients are not properly assessed and addressed. Patients with advanced colorectal cancer can face unique challenges that are stoma- or bowel-related in addition to other symptom burden such as pain, fatigue, and existential distress that have deleterious consequences on their psychological and social functioning. This pilot study aims to test an intervention for patients specifically with advanced colorectal cancer that incorporates culturally-appropriate topics. Using a randomized selection design, we will investigate the feasibility and acceptability of the intervention and obtain an initial estimate of efficacy of the intervention. This pilot study will yield useful information to inform the preparation of a larger, phase III confirmatory study.

DETAILED DESCRIPTION:
Cancer is the leading cause of death in Singapore and colorectal cancer is the most frequently diagnosed cancer in males and second most frequently diagnosed cancer in females, accounting for 17% and 13% of all cancers respectively. Such high incidence rates are consistent with reports of colorectal cancer being a disease of ageing and developed nations . A total of 8931 new cases of colorectal cancer were diagnosed in Singapore from 2009 and 2013, with data indicating a steep increase in incidence rate for patients aged 50 and above. Given that the number of adults aged 65 years and older to double from 2009 to 2030 (Singapore Department of Statistics), the number of colorectal cancer cases are also expected to increase.

Advanced colorectal cancer refers to stage IV cancer of the colon or rectum that cannot be cured and has metastasized to at least one distant organ or set of lymph nodes, and that will likely continue to spread, leading to end of life (National Cancer Institute). In Singapore between 2009 and 2013, approximately 25% of colorectal cancer cases were at stage IV. According to the U.S. NCI's SEER database of patients from 2004-2010, 5-year survival rates for stage IV colon and rectal cancer were 11% and 12% respectively, suggesting these patients are or will soon be managing symptoms of their disease like pain while psychologically confronting end-of-life.

The news of metastatic disease, treatment failure, and/or bleak prognosis can be demoralizing for some patients and characterized by shock, denial, anger, anxiety, and depression which can interfere with everyday living. Studies have reported about one-third to half of advanced cancer patients experience psychological distress and existential crises, yet studies indicate the needs of these patients are not properly assessed and addressed as healthcare providers tend to focus more on patients' physical problems and do not have the time and perceived competency to address emotional distress.

Colorectal cancer comes with its own set of challenges that can significantly alter patients' daily living and affect patient psychological well-being and quality of life. Bowel-related issues have been reported to present physical, psychological, and social challenges to patients and survivors. For instance, patients with surgically-created stoma as part of treatment may face complications of leakage, skin, and odour issues that can lead to anxiety, disturbance in body image, low self-esteem, and social isolation. Furthermore, clinical anecdotes have pointed toward this patient population being concerned about lifestyle factors influencing their disease progression, especially diet. Psychological care has been increasingly recognized as an important part of treatment for this population at such a vulnerable time. Psychological care aims to address patients' mood and worries as they deal with their illness and to help patients find a sense of meaning in their life despite their cancer-related suffering. Unfortunately, psychological care as part of oncology supportive/ palliative services is still very rudimentary in Singapore.

Cognitive behavioural therapy is a widely used, evidence-based therapy that focuses on cognitions, emotions, and behaviour change to address patient distress. This framework has been successfully applied in the treatment of many disorders, including anxiety disorders, depression, chronic pain, and insomnia. It is posited that psycho-behavioural interventions (PBIs) that are based on cognitive-behavioural frameworks can be designed to meet the needs of cancer patients by targeting and modifying their maladaptive thoughts about the disease and treatment (e.g., irrational beliefs, negative attitudes, unrealistic expectations) and their behaviour (e.g., maladaptive coping strategies, isolation, self-negligence). This can be done by teaching patients strategies such as cognitive restructuring, meaning-making, relaxation, activity-pacing, effective communication with others, and utilization of social support. By learning these skills, patients are expected to have increased health-related self-efficacy (i.e., belief in the capacity to manage one's health) that may act as a buffer from them prematurely adopting the "sick role". Self-efficacy can be extremely important in the context of advanced cancer as it allows patients to feel more in control of a situation that is often distressing because of the uncertainty associated with the illness. This in turn may have an effect on patient psychological well-being, symptom management, and utilization of healthcare services such as emergency department (ED) visits and inpatient hospitalizations.

The efficacy of PBIs in alleviating physical symptoms in early-stage cancer has been well-documented. However, the role of such intervention for advanced cancer patients is less clear due to lack of well-designed studies. Advanced disease has unique challenges; for instance, more severe physical symptoms and confrontation of existential meaning as patients approach end of life. This can be associated with greater distress and suffering for patients. A recent review noted that interpretation of the efficacy/effectiveness of PBIs for advanced cancer is limited by the paucity of randomized-controlled studies and lack of racial/ethnic diversity in patients.

The current study aims to investigate the feasibility and acceptability of a PBI designed for advanced colorectal patients implemented in a Singapore context. The intervention will be facilitated by clinical psychologists whose specialty area is psycho-oncology, so as to allow in-depth discussions about suffering associated with cancer and confrontation of end-of-life issues. In this early phase trial, we think it is prudent to conduct the pilot intervention with a homogeneous cancer site so that we can teach symptom management skills that are specific to colorectal cancer. Additionally, we prefer to keep the disease characteristics, prognosis, and indicated treatments as similar as possible across our sample. Such homogeneity prevents the dilution of the intervention effects and facilitates the aim of obtaining an initial estimate of intervention efficacy. The intervention will be unique in that it will include a) therapeutic discussion on legacy building as a way to open discussion about fear of death; b) addressing changed family dynamics, which is important in an Asian context, and c) discussing adaptation to living with bowel-related issues that are a common cause of distress for this patient population. It will be important to use a randomized-controlled design, which is the gold-standard, to provide a definitive answer on the role of PBIs for advanced cancer patients.

In summary, the significance of the study is twofold. Firstly, the proposed PBI pilot study will provide essential, useful information on feasibility and acceptability of providing low-cost, psychological care to advanced colorectal cancer patients that have the potential to address their distress and reduce unnecessary healthcare utilization in Singapore. Secondly, this would be an opportunity to add to the larger body of knowledge on the role of PBIs in provision of supportive care in an Asian setting and beyond. The results will be informative in deciding the worthiness of a phase III confirmatory study. Patients require support throughout the course of their cancer treatment, and currently there are gaps in provision of psychological care for patients with advanced cancer in Singapore's healthcare system. Our long-term goal is to implement evidence-based, cost-effective and scalable psychosocial support as a standard part of supportive care in Singapore.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older
2. Diagnosis of stage IV colorectal cancer
3. Able and willing to attend outpatient therapy appointments
4. Speak and read English or Chinese language

Exclusion Criteria:

1. Serious mental illness (e.g., schizophrenia, bipolar disorder) indicated by medical records
2. Visual, hearing, or cognitive impairment that will interfere with intervention
3. Unaware they have cancer

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The feasibility of the intervention will be tested through enrolment rates. | Up to 8 weeks
  Feasibility of the intervention will be assessed through enrolment rates, rejection rates and exclusion rates.
The acceptability of the intervention will be assessed through the Client Satisfaction Questionnaire. | Up to 8 weeks
  Acceptability of the intervention will be assessed through patient's reported satisfaction with the program, There are 12 items measuring the perceived quality of the program, usefulness of the program, satisfaction with the intervention, comfort level in working with a mental healthcare provider, likelihood of recommending the intervention to others. Five-point Likert scales will be used for the measurement.

SECONDARY OUTCOMES:
Psychological distress will be accessed through The Hospital Anxiety and Depression Scale (HADS) | Up to 8 weeks
  The Hospital Anxiety and Depression Scale (HADS)(Zigmond & Snaith, 1983) will be used to measure psychological distress. There are 7 items measuring anxiety symptoms (HADS-A) and 7 items measuring depressive symptoms (HADS-D). An overall HADS score representing psychological distress will be calculated. This measure has been translated into Singaporean Mandarin and validated for use in Singapore.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Teo, Ph.D., Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National Cancer Centre, Singapore, Singapore

REFERENCES:
- [Background] Campbell CL, Campbell LC. A systematic review of cognitive behavioral interventions in advanced cancer. Patient Educ Couns. 2012 Oct;89(1):15-24. doi: 10.1016/j.pec.2012.06.019. Epub 2012 Jul 12. PMID 22796302
- [Background] Tan PY, Tien Tau LC, Lai Meng OY. Living With Cancer Alone? The Experiences of Singles Diagnosed With Colorectal Cancer. J Psychosoc Oncol. 2015;33(4):354-76. doi: 10.1080/07347332.2015.1045678. PMID 25996668
- [Background] Zhang M, Chan SW, You L, Wen Y, Peng L, Liu W, Zheng M. The effectiveness of a self-efficacy-enhancing intervention for Chinese patients with colorectal cancer: a randomized controlled trial with 6-month follow up. Int J Nurs Stud. 2014 Aug;51(8):1083-92. doi: 10.1016/j.ijnurstu.2013.12.005. Epub 2013 Dec 17. PMID 24406033
- [Background] Sanson-Fisher R, Girgis A, Boyes A, Bonevski B, Burton L, Cook P. The unmet supportive care needs of patients with cancer. Supportive Care Review Group. Cancer. 2000 Jan 1;88(1):226-37. doi: 10.1002/(sici)1097-0142(20000101)88:13.3.co;2-g. PMID 10618627